CLINICAL TRIAL: NCT03078452
Title: Comparison of Quality of Bone Marrow Biopsy and Patient Convenience and Pain Control by a Battery Powered Drill Versus Conventional Methods in Patients With Plasma Cell Disorders
Brief Title: Evaluating Effectiveness of Powered Drill Bone Marrow Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00075658; NCI-2017-00308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship2656-14 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-03-13 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (biopsy using power drill) (Experimental): Patients undergo bone marrow biopsy using the power drill. Patients complete questionnaires at baseline, 30 minutes after biopsy, and on days 1, 3, and 7.
  Interventions: Device: Power drill
- Arm II (biopsy using Jamshidi needle) (Active Comparator): Patients undergo bone marrow biopsy using the traditional Jamshidi needle. Patients complete questionnaires at baseline, 30 minutes after biopsy, and on days 1, 3, and 7.
  Interventions: Device: Jamshidi needle

INTERVENTIONS:
Device: Power drill — Undergo bone marrow biopsy using power drill
  Arms: Arm I (biopsy using power drill)
Device: Jamshidi needle — Undergo bone marrow biopsy using Jamshidi needle
  Arms: Arm II (biopsy using Jamshidi needle)

SUMMARY:
Since the introduction of the Jamshidi needle in 1971, new advances in bone marrow sampling have not been seen. In 2007, a new battery-powered bone marrow biopsy system was developed. This technology, using a battery-powered drill to operate the needle accessing the posterior iliac bone, was approved by the Food and Drug Administration (FDA) and is currently commercially available.

Few randomized controlled trials (RCTs) have compared the use of the battery-powered bone marrow biopsy system to the Jamshidi needle (the traditional manual) method of bone marrow sampling. This research study is designed to evaluate the effectiveness of the Jamshidi needle compared to the battery-powered bone marrow biopsy system.

100 participants will be enrolled in this study at Emory University.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assessing the quality and quantity of bone marrow core biopsies.

SECONDARY OBJECTIVES:

I. Assessing the nature of pain by established visual analogue scale (VAS) questionnaires.

II. Timing of the actual procedure.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo bone marrow biopsy using the power drill.

ARM II: Patients undergo bone marrow biopsy using the traditional Jamshidi needle.

All patients complete questionnaires at baseline, 30 minutes after biopsy, and on days 1, 3, and 7.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* All patients with existing plasma cell disorders and no history of psychiatric disorders who can receive conscious sedation are eligible to participate in the trial

Exclusion Criteria:

* Pregnant women are excluded from participating in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Nooka, MD, MPH, Principal Investigator — Emory University/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Biopsy Using Power Drill) | Arm II (Biopsy Using Jamshidi Needle)
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Biopsy Using Power Drill) | Arm II (Biopsy Using Jamshidi Needle) | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years] | 65.5 [37 to 79] | 63 [35 to 81] | 64.25 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 49 | 98
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 20 | 34
  White | 36 | 30 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Prior Bone Marrow Aspiration & Biopsies (BMA&B) within the last 2 years [Count of Participants; unit: Participants] | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Bone Marrow Core Biopsy Length (in mm) and Artifacts Assessed by the Pathologist
Description: Bone marrow biopsy length is studied with mean, median, range, and standard deviation and compared by two-sample t-test.
Time Frame: At the time of biopsy
Measure: Mean (95% Confidence Interval); unit: Millimeters
Arm/Group | Arm I (Biopsy Using Power Drill) | Arm II (Biopsy Using Jamshidi Needle)
Number analyzed (Participants) | 50 | 50
Millimeters | 14 [5 to 30] | 9.5 [3 to 23]

2. Secondary Outcome: Intensity of Pain Measured Using Visual Analogue Scale (VAS) Pain Questionnaire
Description: The VAS (visual analogue scale) for pain is on a 10 point scale. Pain is studied with chi-square, Mann Whitney U test, or Fisher's exact test.
  The pain scale used was 0-10, with 0 being no pain and 10 being the worst pain.
Time Frame: At the time of, 30 minutes, 1, 3, and 7 days after biopsy
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Biopsy Using Power Drill) | Arm II (Biopsy Using Jamshidi Needle)
Number analyzed (Participants) | 50 | 50
score on a scale
  30 minutes | .66 [0 to 6] | .84 [0 to 8]
  1 day after biopsy | 1.62 [0 to 10] | 1.62 [0 to 10]
  3 days after biopsy | .89 [0 to 8] | .63 [0 to 5]
  7 days after biopsy | .18 [0 to 5] | .26 [0 to 5]

3. Secondary Outcome: Time Taken by the Procedure Measured in Seconds Using a Stopwatch
Description: Staff members will use a stopwatch from the beginning to the completion of the procedure (skin to skin). Time taken for procedure is studied with mean, median, range, and standard deviation and compared by two-sample t-test.
Time Frame: At the time of biopsy
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Arm I (Biopsy Using Power Drill) | Arm II (Biopsy Using Jamshidi Needle)
Number analyzed (Participants) | 50 | 50
Seconds | 7 [3 to 24] | 10.5 [4 to 30]

ADVERSE EVENTS:
Time Frame: Collected for each patient through day +7 after enrollment
Arm/Group | Arm I (Biopsy Using Power Drill) | Arm II (Biopsy Using Jamshidi Needle)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03078452/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03078452/ICF_001.pdf